CLINICAL TRIAL: NCT07305558
Title: Ultrasound Guided Microdochectomy in Chronic Non Dilated Single Duct Nipple Discharge
Brief Title: Microdochectomy for Chronic Non Dilated Single Duct Nipple Discharge
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, lecturer of general surgery, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1248\27-4-2025
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Nipple Discharge
Keywords: nipple discharge; microdochectomy; breast
MeSH Terms: conditions — Galactorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with single milk duct discharge (Experimental)
  Interventions: Procedure: ultrasound guided microdochectomy

INTERVENTIONS:
Procedure: ultrasound guided microdochectomy — ultrasound was used to perform microdochectomy for single not dilated milk duct without cannulation

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of a new technique in treatment of single milk duct discharge. The main questions it aims to answer are:

Does ultrasound guided microdochectomy is feasible in non dilated milk duct? What are the surgical outcomes of this technique?

Participants will:

Had ultrasound microdochectomy After discharge, patients will visit the clinic twice every week for two weeks, a visit or call after 3 month

ELIGIBILITY:
Inclusion Criteria:

* females above 18 years old with single not dilated milk duct discharge after failure of medical treatment

Exclusion Criteria:

* breast cancer
* patients with multiple or dilated milk duct discharge.
* contraindications to surgery or ‬anaesthesia
* patient above 18 years old
* patients refuse to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — this problem is evident only in female breast
Enrollment: 15 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Nipple discharge | from first day after surgery to 3 months after surgery
  stop of spontaneous and induced nipple discharge by absence of stain on dressing and clothes and by squeezing the nipple

SECONDARY OUTCOMES:
operation time | from skin incision to closure
  operation time is calculated in minutes
Bleeding | from skin incision to skin closure
  Bleeding is evaluated in mm using gravimetric and direct vision methods
post operative pain | from the day of surgery to one week after surgery
  post operative pain is assessed using the visual analogue scale. The total score is out of 10 (1 means painless, 10 means painful)
hospital stay | from the first day of surgery to 3 days after surgery
  hospital stay is recorded in days
wound infection | from one day to 2 weeks after surgery
  wound infection diagnosed by direct vision of pus or ultrasound of the breast

CONTACTS AND LOCATIONS:
Overall Officials: Reham Zakaria, M.D, Principal Investigator — faculty of medicine, Zagazig University
Locations (1):
- faculty of medicine, Zagazig University, Zagazig, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
data will be available on demand by direct contact to the principle investigator